CLINICAL TRIAL: NCT01597492
Title: A Phase 4, Multi-Center, Randomized, Open-Label Study to Evaluate the Effect of BENLYSTA™ (Belimumab; HGS1006) on Vaccine Responses in Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: A Study to Evaluate the Effect of Belimumab on Vaccine Responses in Subjects With Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Human Genome Sciences Inc., a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 115470; HGS1006-C1117 (Other: Human Genome Sciences Inc.)
Record Dates: First submitted 2012-05-08; First posted 2012-05-14 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Antibodies; Vaccines; SLE; Immune System Diseases; Biological Therapy; Autoimmune Diseases; Pneumococcal Vaccines; Lupus; Immunoglobulins; Vaccination; Belimumab; Biological Agents; Immunization
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Immune System Diseases; Autoimmune Diseases | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Belimumab plus Early Vaccination (Experimental): Belimumab plus Early Vaccination
  Interventions: Biological: Belimumab plus Early Vaccination
- Belimumab plus Late Vaccination (Experimental): Belimumab plus Late Vaccination
  Interventions: Biological: Belimumab plus Late Vaccination

INTERVENTIONS:
Biological: Belimumab plus Early Vaccination — Belimumab 10 mg/kg IV plus standard therapy for SLE is administered on Days 28, 42, 56, and every 28 days thereafter through Week 32 (9 doses). Pneumococcal vaccination is administered 4 weeks prior to the first dose of belimumab.
  Other Names: BENLYSTA™
  Arms: Belimumab plus Early Vaccination
Biological: Belimumab plus Late Vaccination — Belimumab 10 mg/kg IV plus standard therapy for SLE is administered on Days 0, 14, 28, and then every 28 days thereafter through Week 28 (9 doses). Pneumococcal vaccination is administered 24 weeks after the first dose of belimumab.
  Other Names: BENLYSTA™
  Arms: Belimumab plus Late Vaccination

SUMMARY:
The purpose of this study is to assess the impact of belimumab on immune response to pneumococcal vaccine in subjects with Systemic Lupus Erythematosus (SLE).

DETAILED DESCRIPTION:
All patients in this study will receive belimumab plus standard therapy for SLE and vaccination against pneumococcus. Patients will be randomized to receive pneumococcal vaccination either 4 weeks prior (early vaccination group) or 24 weeks after (late vaccination group) their first belimumab dose. Vaccine response will be assessed 4 weeks after vaccine administration.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of SLE by American College of Rheumatology (ACR) criteria.
* Active SLE disease.
* Autoantibody-positive.
* Have antibodies with titers >1.0 microgram (mcg)/mL to no more than 9 of the 23 serotypes present in the pneumococcal vaccine.
* Have the ability to understand the requirements of the study, provide written informed consent, and comply with the study protocol procedures.

Key Exclusion Criteria:

* Pregnant or nursing.
* Have received any prior treatment with belimumab.
* Have received a live vaccine within the past 30 days.
* Have received a pneumococcal vaccination with the past 5 years.
* Have a history of severe allergic reaction to a vaccine, contrast agents (such as those used for x-rays and CT scans), or biological medicines.
* Have required management of an infection or have had infections that keep coming back within the past 60 days.
* Hepatitis B: Serologic evidence of Hepatitis B (HB) infection based on the results of testing for HB surface antigen (HBsAg) and anti-HB core antibody (anti-HBc):

  * Subjects positive for HBsAg are excluded.
  * Subjects negative for HBsAg but positive for anti-HBc, regardless of anti-HBs antibody status, are excluded.
* Hepatitis C: Positive test for Hepatitis C antibody.
* Known human immunodeficiency virus (HIV) infection.
* Have current drug or alcohol abuse or dependence.
* Have a Grade 3/4 immunoglobulin (Ig)G deficiency (IgG level <400 milligrams [mg]/ deciliter [dL]) or IgA deficiency (IgA level <10 mg/dL).
* Subjects who have evidence of serious suicide risk including any history of suicidal behavior in the last 6 months and/or suicidal ideation with some intent to act in the last 2 months or who in the investigator's judgment, pose a significant suicide risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-05-31 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- United States (14):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Paradise Valley, Arizona
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Cumberland, Maryland
  - GSK Investigational Site, Hagerstown, Maryland
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Burlington, Vermont
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Azoicai T, Antoniu S, Caruntu ID, Azoicai D, Antohe I, Gavrilovici C. Belimumab and antipneumococcal vaccination in patients with systemic lupus erythematosus. Expert Rev Clin Immunol. 2018 Mar;14(3):175-177. doi: 10.1080/1744666X.2018.1429269. Epub 2018 Jan 22. PMID 29336179
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants with systemic lupus erythematosus (SLE) were randomized in 7:9 ratio to receive pneumonococcal vaccination either 4 weeks prior (early cohort) or 24 weeks after (late cohort) their first belimumab dose of 10 milligram (mg)/kilogram (kg) intravenously (IV).
Pre-assignment Details: A total of 79 participants were enrolled, of which 34 were randomised to the early cohort and 45 were randomized to the late cohort. All randomized participants received at least 1 dose of vaccine and/or belimumab and were included in the Intent-to-Treat (ITT) Population.
Groups:
- Belimumab Plus Early Vaccination: Participants received pneumococcal vaccination on Day 0, 4 weeks prior to the first dose of belimumab. Open-label belimumab 10 mg/kg IV was dosed on Days 28, 42, 56, and every 28 days thereafter until Week 32 (a total of 9 doses) plus standard therapy for SLE.
- Belimumab Plus Late Vaccination: Participants received pneumococcal vaccination on Day 168 (Week 24). Open-label belimumab 10 mg/kg IV was dosed on Days 0, 14, 28, and every 28 days thereafter until Week 28 (a total of 9 doses) plus standard therapy for SLE.
Period: Overall Study
Arm/Group | Belimumab Plus Early Vaccination | Belimumab Plus Late Vaccination
Started | 34 | 45
Completed | 28 | 41
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Other Reason | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belimumab Plus Early Vaccination | Belimumab Plus Late Vaccination | Total
Number analyzed (Participants) | 34 | 45 | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.0 (12.57) | 38.6 (12.31) | 39.6 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 43 | 72
  Male | 5 | 2 | 7
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 25 | 27 | 52
  Black or African American | 8 | 12 | 20
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Mixed Race | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Antibody Responses to at Least One of the 23 Pneumococcal Vaccine Serotypes 4 Weeks Post-vaccination
Description: A positive immune response to at least one pneumococcal serotype is defined as a 2-fold or greater increase from pre-vaccination levels. For unquantifiable pre-vaccination antibody levels, a positive antibody response was considered as a post-vaccination level >=0.6 micrograms (µg)/milliliter (mL). Post-vaccination pneumococcal titers were assessed on Day 28 (Week 4) prior to the first dose of belimumab in the early cohort and on Day 196 (Week 28) prior to the last belimumab dose in the late cohort. Evaluable participants for the early cohort included those who received the vaccination at Day 0 and had titers drawn at Week 4. For the late cohort, evaluable participants received at least 5 of the 7 doses of belimumab up through Week 24, received the vaccination at Week 24, and had titers drawn at Week 28.
Time Frame: Four weeks after vaccination
Population: As-treated Population: all participants who received at least one dose of belimumab. All analyses of vaccine titers were performed on the As-treated Population.
Measure: Number; unit: Participants
Arm/Group | Belimumab Plus Early Vaccination | Belimumab Plus Late Vaccination
Number analyzed (Participants) | 33 | 41
Participants | 32 | 40

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until follow-up (up to 8 weeks following administration of the last dose of belimumab).
Description: SAEs and non-serious AEs were reported for the ITT population, comprised of participants who were randomized to treatment, and received at least one dose of study medication. Treatment-emergent AEs were those that occurred on or after the first belimumab infusion, which was Week 4 for the early cohort and Week 0 for the late cohort.
Arm/Group | Belimumab Plus Early Vaccination | Belimumab Plus Late Vaccination
Serious Adverse Events (participants affected / at risk) | 4/34 | 3/45
Other Adverse Events (participants affected / at risk) | 21/34 | 32/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab Plus Early Vaccination (N=34) | Belimumab Plus Late Vaccination (N=45)
Any event (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Pericarditis lupus (Cardiac disorders) | 1 | 0
Any event (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Any event (Renal and urinary disorders) | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Glomerulonephritis proliferative (Renal and urinary disorders) | 1 | 0
Any event (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Any event (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Any event (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab Plus Early Vaccination (N=34) | Belimumab Plus Late Vaccination (N=45)
Any event (Infections and infestations) | 10 | 20
Gastroenteritis viral (Infections and infestations) | 1 | 6
Viral upper respiratory tract infection (Infections and infestations) | 3 | 4
Bronchitis bacterial (Infections and infestations) | 2 | 4
Upper respiratory tract infection bacterial (Infections and infestations) | 2 | 3
Sinusitis (Infections and infestations) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 2
Any event (Gastrointestinal disorders) | 7 | 12
Nausea (Gastrointestinal disorders) | 6 | 9
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 1 | 4
Any event (Musculoskeletal and connective tissue disorders) | 6 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Any event (Nervous system disorders) | 5 | 5
Dizziness (Nervous system disorders) | 4 | 2
Headache (Nervous system disorders) | 2 | 3
Any event (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Any event (Psychiatric disorders) | 1 | 4
Depression (Psychiatric disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.